CLINICAL TRIAL: NCT05727046
Title: Investigation of the Usability of the Dynamic Scaffolding System An Adaptive Mobility Device in Children With Special Needs and Parental Satisfaction
Brief Title: Investigation of the Usability of the Dynamic Scaffolding System
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Turgay Altunalan, Principal Investigator, Karadeniz Technical University
Other Study IDs: KaradenizTechnicalU; Beyzanur Dikmen (Other: Uskudar University); Melek Vatansever (Other: Uskudar University)
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Child Development Disorder; Child Development; Assistive Technology
Keywords: children with disability; assistive device; walker; children; Dynamic Scaffolding System; Parental satisfaction
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy and Children with other diagnoses: Of the children with special needs included in the study, 60% were parents of children with cerebral palsy.
  40% of the children with special needs included in the study had Hydrocephalus, Arthrogryposis, Multiplex Congenita, Down Syndrome, Microcephaly, Alpha-thalassemia mental retardation syndrome (ATRX), Spinal Muscular Atrophy (SMA) Type 1, Spinal Muscular Atrophy (SMA) Type 2, L2 hydroxy glutaric aciduria, Prader Willi syndrome, Periventricular leukomalacia grade 1, Hypotonia, Angelman syndrome, Genetic chromosomal abnormality, Dandy-walker syndrome, Western syndrome, Infantile epileptic encephalopathy, Stroke-like migraine attacks after radiation therapy (SMART syndrome), Trigonocephaly, Motor developmental delay, Lissencephaly, Spina bifida, Leigh syndrome and Epilepsy.

SUMMARY:
The aim of the present study was to compare the duration of use of the Dynamic Scaffolding System (DSS) in children with different levels of motor impairment, to report adverse events during use, and to examine parental satisfaction. One hundred children with special needs aged between 9 and 108 months who had used the DSS device for at least 6 months and their parents were included in the study. The duration of daily use of the DSS device by the children, any adverse events during use, and parental satisfaction were assessed using the Quebec 2.0 Assistive Technology User Satisfaction Assessment Questionnaire.

DETAILED DESCRIPTION:
Children with special needs with mobility difficulties use various assistive devices to benefit from the beneficial effects of standing upright and moving. These devices have beneficial effects on improving children's motor skills and increasing their social interaction and participation. In addition, during the use of assistive devices, there are some limitations related to size, weight, usability, mobility, and adaptability to children. Considering these limitations, the Dynamic Scaffolding System (DSS) device was developed. The DSS device aims to position children with moderate to severe mobility impairment vertically (standing and sitting) and to step with support. The aim of the current study was to compare the duration of use of the Dynamic Scaffolding System (DSS) device in children with different levels of motor impairment, to report adverse events during use, and to examine parental satisfaction. One hundred children with special needs (60% cerebral palsy, 40% other diagnoses: genetic, metabolic, neuromuscular diseases) aged between 9 and 108 months (mean 44.94±17.59) and their parents (94% mother, 6% father) who had used the DSS device for at least 6 months were included in the study. Data were collected from the participants via telephone interview. Demographic data such as age, gender, diagnosis, and level of motor impairment were recorded. Children's daily use of the DSS device, any adverse events during use, and parental satisfaction were assessed using the Quebec 2.0 Assistive Technology User Satisfaction Assessment Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children with motor disabilities

Exclusion Criteria:

* If children did not use Dynamic Scaffolding System for less than one month

Ages: 9 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with motor difficulties
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Everyday Usage Time of Dynamic Scaffolding System (DSS) | After 1 months experience of Dynamic Scaffolding System
  Dynamic Scaffolding System is an assistive device for children with special needs. We measure the usage time of DSS by the chronometer.

SECONDARY OUTCOMES:
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | After 1 months experience of Dynamic Scaffolding System
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components such as Devices and Services. Psychometric properties have been tested with respect to test-retest stability. The participants give answers on a 5-point Likert Scale. The high point means better results.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Uskudar University, Istanbul
  - Karadeniz Technical University, Trabzon

IPD SHARING:
Plan to Share IPD: No